CLINICAL TRIAL: NCT04401176
Title: A Randomized Trial of Bladder Instillations Versus Onabotulinumtoxin A for Treatment of Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Bladder Instillations Versus Onabotulinumtoxin A for Treatment of Interstitial Cystitis/Bladder Pain Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKW_01-2020
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Heparin; onabotulinum toxin A

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Heparin & Alkalinized Lidocaine Bladder Instillation (Active Comparator): Six weekly bladder instillations, each instillation consisting of 40,000 IU Heparin, 200mg lidocaine, 2ml 8.4% sodium bicarbonate, sterile water for a total volume 50 milliliters (mL).
  Interventions: Drug: Heparin & Alkalinized Lidocaine Bladder Instillation
- Intradetrusor Onabotulinumtoxin A Injection (Active Comparator): 100 units onabotulinumtoxinA reconstituted in 10mL of injectable saline, injected in 20 sites with 0.5mL per injection along the posterior wall of the bladder above the trigone.
  Interventions: Drug: Onabotulinum Toxin A

INTERVENTIONS:
Drug: Heparin & Alkalinized Lidocaine Bladder Instillation — Bladder instillation instilled via catheter and to dwell for minimum of 30 minutes prior to spontaneous void
  Arms: Heparin & Alkalinized Lidocaine Bladder Instillation
Drug: Onabotulinum Toxin A — Intradetrusor onabotulinumtoxinA injection (0.5mL x 20 sites)
  Arms: Intradetrusor Onabotulinumtoxin A Injection

SUMMARY:
Recognition of interstitial cystitis (IC)/bladder pain syndrome (BPS) is increasing. There is a dire need to develop effective treatment options for these patients as it manifests as more than a physical disease, affecting general and psychological health as well. Existing trials comparing varying bladder instillation formulations have not identified an optimal bladder instillation therapy, however existing studies support combined heparin and alkalinized lidocaine bladder instillation as an affordable and effective treatment for IC/BPS. Additionally, intradetrusor onabotulinumtoxinA injection has been well established for the treatment of overactive bladder (OAB), a constellation of symptoms similar to that of IC/BPS. OnabotulinumtoxinA has now come into the forefront for treatment of OAB due to its efficacy, safety profile, and absence of cognitive effects related to the previous mainstay anticholinergic treatment. While both bladder instillation and onabotulinumtoxinA therapy have been shown to be effective for treatment of IC/BPS, a direct comparison of these treatments has not been performed. We therefore designed a randomized controlled trial to compare the efficacy of heparin with alkalized local anesthetic bladder instillation versus intradetrusor onabotulinumtoxinA injection in treating IC/BPS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥ 18 years of age
* O'Leary-Sant questionnaire score ≥ 6
* Ability to follow study instructions and complete all required follow-up

Exclusion Criteria:

* Contraindications and/or allergies to medications used
* Known alternative diagnosis explaining bladder pain symptoms
* Bladder instillation within the past 3 months
* Intradetrusor onabotulinumtoxinA injection within the past 6 months
* Use of ≥ 400 units of onabotulinumtoxinA in the last 3 months
* Inability or unwillingness to self-catheterize
* Post-void residual > 200mL
* Concurrent procedural treatment (including hydrodistension, sacral neuromodulation)
* Current use of vaginal pessary/devices
* Untreated symptomatic prolapse > pelvic organ prolapse quantification system (POP-Q) stage 2
* Females who are pregnant or planning a pregnancy during the study or who think that they may be pregnant at the start of the study and who are unwilling or unable to use a reliable form of contraception during the study
* Inability to speak/read English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in O'Leary-Sant questionnaire scores from baseline between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | Baseline, 8-10 weeks
  Consists of O'Leary-Sant Symptom and Problem Index, total score 0-36.

SECONDARY OUTCOMES:
Change in O'Leary-Sant questionnaire scores from baseline between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | Baseline, 4-6 weeks, 6-9 months
  Consists of O'Leary-Sant Symptom and Problem Index. Total score 0-36
Change in pain scores using the Defense and Veterans Pain Rating Scale (visual analog scale) between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | Baseline, 4-6 weeks, 8-10 weeks, 6-9 months
  Scale of 0-10 (0= no pain, 10 = worst pain)
Change in Female Sexual Function Index (FSFI) score between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | Baseline, 4-6 weeks, 8-10 weeks
  FSFI evaluates 5 domains of female sexual function including desire, arousal, lubrication, orgasm, satisfaction, and pain. Total score 2-36.
Change in Female Sexual Distress Scale-Revised (FSDS-R) score between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | Baseline, 4-6 weeks, 8-10 weeks
  FSDS-R evaluates distress associated with inadequate/impaired sexual function. Total score 0-52.
Change in 12-item Short Form Survey (SF-12) score between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | Baseline, 4-6 weeks, 8-10 weeks
  SF-12 is a general health questionnaire that evaluates quality of life measures, divided into mental and physical component scores.
Change in bladder capacity between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | Baseline, 4-6 weeks, 8-10 weeks
  Bladder capacity via 1-day bladder diary
Incidence of adverse outcomes between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | 8-10 weeks
  Adverse outcomes to be defined specific to medication administered (urinary tract infection in both bladder instillation and onabotulinumtoxinA injection groups, urinary retention requiring catheterization, systemic effects related to onabotulinumtoxinA group only)
Patient perceptions of treatment between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | 6-9 months
  "How convenient or inconvenient was it to follow the treatment schedule as instructed?" (Scale 1-5 extremely inconvenient - extremely convenient) "How satisfied or dissatisfied are you in the ability of the treatment to treat your condition?" (Scale 1-5 extremely dissatisfied - extremely satisfied) "Taking all things into account, how satisfied or dissatisfied are you with this treatment?" (Scale 1-5 extremely dissatisfied - extremely satisfied) "How willing would you be to undergo this treatment again?" (Scale 1-5 extremely unwilling - extremely willing).
Incidence of re-treatment between bladder instillation and intradetrusor onabotulinumtoxinA injection groups | 6-9 months
  Re-treatment defined as additional course or crossover treatment outside of assigned treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hanno P, Dmochowski R. Status of international consensus on interstitial cystitis/bladder pain syndrome/painful bladder syndrome: 2008 snapshot. Neurourol Urodyn. 2009;28(4):274-86. doi: 10.1002/nau.20687. PMID 19260081
- [Background] Berry SH, Elliott MN, Suttorp M, Bogart LM, Stoto MA, Eggers P, Nyberg L, Clemens JQ. Prevalence of symptoms of bladder pain syndrome/interstitial cystitis among adult females in the United States. J Urol. 2011 Aug;186(2):540-4. doi: 10.1016/j.juro.2011.03.132. Epub 2011 Jun 16. PMID 21683389
- [Background] Clemens JQ, Link CL, Eggers PW, Kusek JW, Nyberg LM Jr, McKinlay JB; BACH Survey Investigators. Prevalence of painful bladder symptoms and effect on quality of life in black, Hispanic and white men and women. J Urol. 2007 Apr;177(4):1390-4. doi: 10.1016/j.juro.2006.11.084. PMID 17382739
- [Background] Rothrock NE, Lutgendorf SK, Hoffman A, Kreder KJ. Depressive symptoms and quality of life in patients with interstitial cystitis. J Urol. 2002 Apr;167(4):1763-7. PMID 11912405
- [Background] Rothrock N, Lutgendorf SK, Kreder KJ. Coping strategies in patients with interstitial cystitis: relationships with quality of life and depression. J Urol. 2003 Jan;169(1):233-6. doi: 10.1016/S0022-5347(05)64075-X. PMID 12478143
- [Background] Nickel JC, Payne CK, Forrest J, Parsons CL, Wan GJ, Xiao X. The relationship among symptoms, sleep disturbances and quality of life in patients with interstitial cystitis. J Urol. 2009 Jun;181(6):2555-61. doi: 10.1016/j.juro.2009.02.030. Epub 2009 Apr 16. PMID 19375108
- [Background] Nickel JC, Tripp DA, Pontari M, Moldwin R, Mayer R, Carr LK, Doggweiler R, Yang CC, Mishra N, Nordling J. Psychosocial phenotyping in women with interstitial cystitis/painful bladder syndrome: a case control study. J Urol. 2010 Jan;183(1):167-72. doi: 10.1016/j.juro.2009.08.133. PMID 19913812
- [Background] Payne CK, Joyce GF, Wise M, Clemens JQ; Urologic Diseases in America Project. Interstitial cystitis and painful bladder syndrome. J Urol. 2007 Jun;177(6):2042-9. doi: 10.1016/j.juro.2007.01.124. PMID 17509284
- [Background] Hurst RE. Structure, function, and pathology of proteoglycans and glycosaminoglycans in the urinary tract. World J Urol. 1994;12(1):3-10. doi: 10.1007/BF00182044. PMID 8012413
- [Background] Parsons CL. The role of the urinary epithelium in the pathogenesis of interstitial cystitis/prostatitis/urethritis. Urology. 2007 Apr;69(4 Suppl):9-16. doi: 10.1016/j.urology.2006.03.084. PMID 17462486
- [Background] Cvach K, Rosamilia A. Review of intravesical therapies for bladder pain syndrome/interstitial cystitis. Transl Androl Urol. 2015 Dec;4(6):629-37. doi: 10.3978/j.issn.2223-4683.2015.10.07. PMID 26816864
- [Background] Basbaum AI, Bautista DM, Scherrer G, Julius D. Cellular and molecular mechanisms of pain. Cell. 2009 Oct 16;139(2):267-84. doi: 10.1016/j.cell.2009.09.028. PMID 19837031
- [Background] Henry RA, Morales A, Cahill CM. Beyond a Simple Anesthetic Effect: Lidocaine in the Diagnosis and Treatment of Interstitial Cystitis/bladder Pain Syndrome. Urology. 2015 May;85(5):1025-1033. doi: 10.1016/j.urology.2015.01.021. PMID 25917728
- [Background] Nickel JC, Stephens A, Landis JR, Mullins C, van Bokhoven A, Lucia MS, Ehrlich GD; MAPP Research Network. Assessment of the Lower Urinary Tract Microbiota during Symptom Flare in Women with Urologic Chronic Pelvic Pain Syndrome: A MAPP Network Study. J Urol. 2016 Feb;195(2):356-62. doi: 10.1016/j.juro.2015.09.075. Epub 2015 Sep 26. PMID 26410734
- [Background] Pearce MM, Zilliox MJ, Rosenfeld AB, Thomas-White KJ, Richter HE, Nager CW, Visco AG, Nygaard IE, Barber MD, Schaffer J, Moalli P, Sung VW, Smith AL, Rogers R, Nolen TL, Wallace D, Meikle SF, Gai X, Wolfe AJ, Brubaker L; Pelvic Floor Disorders Network. The female urinary microbiome in urgency urinary incontinence. Am J Obstet Gynecol. 2015 Sep;213(3):347.e1-11. doi: 10.1016/j.ajog.2015.07.009. Epub 2015 Jul 23. PMID 26210757
- [Background] Abernethy MG, Rosenfeld A, White JR, Mueller MG, Lewicky-Gaupp C, Kenton K. Urinary Microbiome and Cytokine Levels in Women With Interstitial Cystitis. Obstet Gynecol. 2017 Mar;129(3):500-506. doi: 10.1097/AOG.0000000000001892. PMID 28178051
- [Background] Nickel JC, Stephens-Shields AJ, Landis JR, Mullins C, van Bokhoven A, Lucia MS, Henderson JP, Sen B, Krol JE, Ehrlich GD; MAPP Research Network. A Culture-Independent Analysis of the Microbiota of Female Interstitial Cystitis/Bladder Pain Syndrome Participants in the MAPP Research Network. J Clin Med. 2019 Mar 26;8(3):415. doi: 10.3390/jcm8030415. PMID 30917614
- [Background] Meriwether KV, Lei Z, Singh R, Gaskins J, Hobson DTG, Jala V. The Vaginal and Urinary Microbiomes in Premenopausal Women With Interstitial Cystitis/Bladder Pain Syndrome as Compared to Unaffected Controls: A Pilot Cross-Sectional Study. Front Cell Infect Microbiol. 2019 Apr 8;9:92. doi: 10.3389/fcimb.2019.00092. eCollection 2019. PMID 31024861
- [Background] Wolfe AJ, Toh E, Shibata N, Rong R, Kenton K, Fitzgerald M, Mueller ER, Schreckenberger P, Dong Q, Nelson DE, Brubaker L. Evidence of uncultivated bacteria in the adult female bladder. J Clin Microbiol. 2012 Apr;50(4):1376-83. doi: 10.1128/JCM.05852-11. Epub 2012 Jan 25. PMID 22278835
- [Background] Weiss JM. Pelvic floor myofascial trigger points: manual therapy for interstitial cystitis and the urgency-frequency syndrome. J Urol. 2001 Dec;166(6):2226-31. doi: 10.1016/s0022-5347(05)65539-5. PMID 11696740
- [Background] Bedaiwy MA, Patterson B, Mahajan S. Prevalence of myofascial chronic pelvic pain and the effectiveness of pelvic floor physical therapy. J Reprod Med. 2013 Nov-Dec;58(11-12):504-10. PMID 24568045
- [Background] Sant GR, Propert KJ, Hanno PM, Burks D, Culkin D, Diokno AC, Hardy C, Landis JR, Mayer R, Madigan R, Messing EM, Peters K, Theoharides TC, Warren J, Wein AJ, Steers W, Kusek JW, Nyberg LM; Interstitial Cystitis Clinical Trials Group. A pilot clinical trial of oral pentosan polysulfate and oral hydroxyzine in patients with interstitial cystitis. J Urol. 2003 Sep;170(3):810-5. doi: 10.1097/01.ju.0000083020.06212.3d. PMID 12913705
- [Background] Foster HE Jr, Hanno PM, Nickel JC, Payne CK, Mayer RD, Burks DA, Yang CC, Chai TC, Kreder KJ, Peters KM, Lukacz ES, FitzGerald MP, Cen L, Landis JR, Propert KJ, Yang W, Kusek JW, Nyberg LM; Interstitial Cystitis Collaborative Research Network. Effect of amitriptyline on symptoms in treatment naive patients with interstitial cystitis/painful bladder syndrome. J Urol. 2010 May;183(5):1853-8. doi: 10.1016/j.juro.2009.12.106. Epub 2010 Mar 29. PMID 20303115
- [Background] Cassinelli G, Naggi A. Old and new applications of non-anticoagulant heparin. Int J Cardiol. 2016 Jun;212 Suppl 1:S14-21. doi: 10.1016/S0167-5273(16)12004-2. PMID 27264866
- [Background] Nickel JC, Moldwin R, Lee S, Davis EL, Henry RA, Wyllie MG. Intravesical alkalinized lidocaine (PSD597) offers sustained relief from symptoms of interstitial cystitis and painful bladder syndrome. BJU Int. 2009 Apr;103(7):910-8. doi: 10.1111/j.1464-410X.2008.08162.x. Epub 2008 Nov 13. PMID 19021619
- [Background] Kuo HC. Urodynamic results of intravesical heparin therapy for women with frequency urgency syndrome and interstitial cystitis. J Formos Med Assoc. 2001 May;100(5):309-14. PMID 11432309
- [Background] Henry R, Patterson L, Avery N, Tanzola R, Tod D, Hunter D, Nickel JC, Morales A. Absorption of alkalized intravesical lidocaine in normal and inflamed bladders: a simple method for improving bladder anesthesia. J Urol. 2001 Jun;165(6 Pt 1):1900-3. doi: 10.1097/00005392-200106000-00014. PMID 11371877
- [Background] Birch BR, Miller RA. Absorption characteristics of lignocaine following intravesical instillation. Scand J Urol Nephrol. 1994 Dec;28(4):359-64. doi: 10.3109/00365599409180513. PMID 7886411
- [Background] Parsons CL, Zupkas P, Proctor J, Koziol J, Franklin A, Giesing D, Davis E, Lakin CM, Kahn BS, Garner WJ. Alkalinized lidocaine and heparin provide immediate relief of pain and urgency in patients with interstitial cystitis. J Sex Med. 2012 Jan;9(1):207-12. doi: 10.1111/j.1743-6109.2011.02542.x. Epub 2011 Nov 14. PMID 22082303
- [Background] Nomiya A, Naruse T, Niimi A, Nishimatsu H, Kume H, Igawa Y, Homma Y. On- and post-treatment symptom relief by repeated instillations of heparin and alkalized lidocaine in interstitial cystitis. Int J Urol. 2013 Nov;20(11):1118-22. doi: 10.1111/iju.12120. Epub 2013 Feb 22. PMID 23432185
- [Background] Davis EL, El Khoudary SR, Talbott EO, Davis J, Regan LJ. Safety and efficacy of the use of intravesical and oral pentosan polysulfate sodium for interstitial cystitis: a randomized double-blind clinical trial. J Urol. 2008 Jan;179(1):177-85. doi: 10.1016/j.juro.2007.08.170. Epub 2007 Nov 14. PMID 18001798
- [Background] Sun Y, Chai TC. Effects of dimethyl sulphoxide and heparin on stretch-activated ATP release by bladder urothelial cells from patients with interstitial cystitis. BJU Int. 2002 Sep;90(4):381-5. doi: 10.1046/j.1464-410x.2002.02912.x. PMID 12175393
- [Background] Shiga KI, Hirano K, Nishimura J, Niiro N, Naito S, Kanaide H. Dimethyl sulphoxide relaxes rabbit detrusor muscle by decreasing the Ca2+ sensitivity of the contractile apparatus. Br J Pharmacol. 2007 Aug;151(7):1014-24. doi: 10.1038/sj.bjp.0707317. Epub 2007 Jun 4. PMID 17549043
- [Background] Perez-Marrero R, Emerson LE, Feltis JT. A controlled study of dimethyl sulfoxide in interstitial cystitis. J Urol. 1988 Jul;140(1):36-9. doi: 10.1016/s0022-5347(17)41478-9. PMID 3288775
- [Background] Rawls WF, Cox L, Rovner ES. Dimethyl sulfoxide (DMSO) as intravesical therapy for interstitial cystitis/bladder pain syndrome: A review. Neurourol Urodyn. 2017 Sep;36(7):1677-1684. doi: 10.1002/nau.23204. Epub 2017 Feb 21. PMID 28220525
- [Background] Erickson DR, Kunselman AR, Bentley CM, Peters KM, Rovner ES, Demers LM, Wheeler MA, Keay SK. Changes in urine markers and symptoms after bladder distention for interstitial cystitis. J Urol. 2007 Feb;177(2):556-60. doi: 10.1016/j.juro.2006.09.029. PMID 17222633
- [Background] Hanno PM, Wein AJ. Conservative therapy of interstitial cystitis. Semin Urol. 1991 May;9(2):143-7. No abstract available. PMID 1712978
- [Background] Kuo HC, Chancellor MB. Comparison of intravesical botulinum toxin type A injections plus hydrodistention with hydrodistention alone for the treatment of refractory interstitial cystitis/painful bladder syndrome. BJU Int. 2009 Sep;104(5):657-61. doi: 10.1111/j.1464-410X.2009.08495.x. Epub 2009 Mar 30. PMID 19338543
- [Background] Welch MJ, Purkiss JR, Foster KA. Sensitivity of embryonic rat dorsal root ganglia neurons to Clostridium botulinum neurotoxins. Toxicon. 2000 Feb;38(2):245-58. doi: 10.1016/s0041-0101(99)00153-1. PMID 10665805
- [Background] Durham PL, Cady R, Cady R. Regulation of calcitonin gene-related peptide secretion from trigeminal nerve cells by botulinum toxin type A: implications for migraine therapy. Headache. 2004 Jan;44(1):35-42; discussion 42-3. doi: 10.1111/j.1526-4610.2004.04007.x. PMID 14979881
- [Background] Liu HT, Kuo HC. Intravesical botulinum toxin A injections plus hydrodistension can reduce nerve growth factor production and control bladder pain in interstitial cystitis. Urology. 2007 Sep;70(3):463-8. doi: 10.1016/j.urology.2007.04.038. PMID 17905097
- [Background] Smith CP, Radziszewski P, Borkowski A, Somogyi GT, Boone TB, Chancellor MB. Botulinum toxin a has antinociceptive effects in treating interstitial cystitis. Urology. 2004 Nov;64(5):871-5; discussion 875. doi: 10.1016/j.urology.2004.06.073. PMID 15533466
- [Background] Giannantoni A, Costantini E, Di Stasi SM, Tascini MC, Bini V, Porena M. Botulinum A toxin intravesical injections in the treatment of painful bladder syndrome: a pilot study. Eur Urol. 2006 Apr;49(4):704-9. doi: 10.1016/j.eururo.2005.12.002. Epub 2006 Jan 4. PMID 16417964
- [Background] Apostolidis A, Dasgupta P, Fowler CJ. Proposed mechanism for the efficacy of injected botulinum toxin in the treatment of human detrusor overactivity. Eur Urol. 2006 Apr;49(4):644-50. doi: 10.1016/j.eururo.2005.12.010. Epub 2006 Jan 4. PMID 16426734
- [Background] Coupland CAC, Hill T, Dening T, Morriss R, Moore M, Hippisley-Cox J. Anticholinergic Drug Exposure and the Risk of Dementia: A Nested Case-Control Study. JAMA Intern Med. 2019 Aug 1;179(8):1084-1093. doi: 10.1001/jamainternmed.2019.0677. PMID 31233095
- See also: American Urological Association Interstitial Cystitis Guidelines — https://www.auanet.org/guidelines/interstitial-cystitis-(ic/bps)-guideline

DOCUMENTS (1):
  • Informed Consent Form (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT04401176/ICF_000.pdf